CLINICAL TRIAL: NCT06897332
Title: Comparing Brain Cortical Activity in Real and Immersive Virtual Reality Manual Dexterity Tasks
Status: Not yet recruiting | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: Real vs iVR Manual Dexterity
Record Dates: First submitted 2025-03-13; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Brain; Virtual Reality; EEG; fNIRS; Manual Dexterity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy individuals
  Interventions: Behavioral: Real-world manual dexterity task; Behavioral: Immersive virtual reality with controllers; Behavioral: Immersive virtual reality with hand-tracking

INTERVENTIONS:
Behavioral: Real-world manual dexterity task — Participants will perform a manual dexterity task involving the displacement of physical cubes
Behavioral: Immersive virtual reality with controllers — Participants will perform a manual dexterity task in an immersive virtual reality environment, requiring them to move virtual cubes using controllers
Behavioral: Immersive virtual reality with hand-tracking — Participants will perform a manual dexterity task in an immersive virtual reality environment, requiring them to move virtual cubes using the hand-tracking technology

SUMMARY:
With advances in technology, virtual reality (VR) is increasingly used in various fields, including rehabilitation, motor learning, and neuroscience. Its ability to provide controlled, immersive, and interactive environments makes it a valuable tool for training and assessment. However, despite its growing adoption, limited evidence exists on how cortical activation in VR compares to real-world conditions. Moreover, brain cortical activity during motor tasks, such as manual dexterity tasks, remains underexplored.

This study aims to compare brain cortical activity in real and immersive virtual reality settings during a manual dexterity task. Secondary objectives include:

* Examining the relationship between brain cortical activity and kinematics in both conditions.
* Comparing brain cortical activity between hand-tracking and controller-based interactions.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Normal-to-corrected vision
* Ability to understand simple instructions

Exclusion Criteria:

* History of seizure
* Recent participation (within the last three months) in a study involving a manual dexterity task in immersive virtual reality
* Neurologic or orthopaedic pathology potentially affecting upper extremity movement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited through word-of-mouth within the Belgian population
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Brain cortical activity | Baseline (at rest: before task performance) and Day 1 (during each of the three task performances within the single study session)
  Measures of brain cortical activity using EEG/fNIRS

SECONDARY OUTCOMES:
Average speed | Day 1 (during each of the three task performances within the single study session)
  Mean instant velocity of the upper extremity during task performance
Maximal movement speed | Day 1 (during each of the three task performances within the single study session)
  Peak instant velocity of the upper extremity during task performance
Movement smoothness | Day 1 (during each of the three task performances within the single study session)
  Spectral arc length of the normalised instant velocity (SPARC) of the upper extremity during task performance
Variation of velocity | Day 1 (during each of the three task performances within the single study session)
  Coefficient of variation of the instant velocity of the upper extremity during task performance
Average distance between thumb and other fingers | Day 1 (during each of the three task performances within the single study session)
  Mean distance between thumb and other fingers during task performance
Variation of distance between thumb and other fingers | Day 1 (during each of the three task performances within the single study session)
  Coefficient of variation of the distance between thumb and other fingers during task performance

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Lejeune, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc UCL
Locations (1):
- Neuro Musculo Skeletal Lab, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No